CLINICAL TRIAL: NCT04894708
Title: Prospective Randomized Study on the Use of Artificial Intelligence (Fujifilm) for Polyp Detection in Colonoscopy
Brief Title: Study on the Use of Artificial Intelligence (Fujifilm) for Polyp Detection in Colonoscopy
Acronym: Fuji AI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: FUJIFILM Deutschland, Branch office of FUJIFILM Europe GmbH (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Thomas Rösch, Director of Department of Interdisciplinary Endoscopy of University Hospital Hamburg Eppendorf, Universitätsklinikum Hamburg-Eppendorf
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PV7284
Record Dates: First submitted 2020-12-01; First posted 2021-05-20 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Screening Colonoscopy; Colonoscopic Control After Polypectomy; Suspected Colon Polyps
MeSH Terms: interventions — Colonoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI colonoscopy (Other): colonoscopy with artificial intelligence added
  Interventions: Procedure: colonoscopy
- conventional colonoscopy (Sham Comparator): conventional colonoscopy
  Interventions: Procedure: colonoscopy

INTERVENTIONS:
Procedure: colonoscopy — addition of polyp detection algorithm by Fujifilm

SUMMARY:
Colonoscopy is currently the best method of detection of intestinal tumors and polyps, particularly because polyps can also be biopsied and removed. There is a clear correlation between the adenoma detection rate and prevented carcinomas, so adenoma detection rate is the main parameter for the outcome quality of diagnostic colonoscopy. The efficiency of preventive colonoscopy needs optimisation by increase in adenoma detection rate, as it is known from many studies that approximately 15-30% of all adenomas can be overlooked. This mainly applies to smaller and flat adenomas. However, since even smaller polyps may be relevant for colorectal cancer development, the aim of colonoscopy should be to preferably be able to recognize all polyps and other changes.The latest and by far the most interesting development in this field is the use of artificial intelligence systems. They consist of a switched-on software with a small computer connected to the endoscope processor; the patient's introduced endoscope is completely unchanged.

The present study therefore compares the adenoma detection rate (ADR) of the latest generation of devices with high-resolution imaging from Fujifilm with and without the connection of artificial intelligence.

DETAILED DESCRIPTION:
Methods of Computer Vision (CV) and Artificial Intelligence (AI) provide completely new opportunities, e.g. in the automatic polyp detection and differentiation of a lesion based on its endoscopic image. Computer vision using artificial intelligence methods means the application of "trained" so-called deep neural net (DNN) with a set of defined images (e.g. everyday scenes) and well-known solutions ( e.g. name of the pictured item; c.f. e.g. the "ImageNet Challenge"). The technical feasibility of using AI algorithms in endoscopy has already been proven in many cases. In the present study, it is an AI system from Fujifilm, which is already clinically usable. By using Fujifilm high-resolution imaging devices in colonoscopies, AI will be added randomly.

ELIGIBILITY:
Inclusion Criteria:

* Persons> 35 years of age who are capable of giving informed consent
* Planned diagnostic colonoscopy (clarification of symptoms, polyp follow-up)
* Screening colonoscopy for men >50 or women > 55 years of age

Exclusion Criteria:

* Colon bleeding
* Colon carcinoma
* Known polyps for removal
* Inflammatory bowel disease
* Colonic stenosis
* Other suspected colon disease for further clarification
* Follow-up care after colon cancer surgery (partial colon resection)
* Anticoagulant drugs that make a biopsy or polypectomy impossible
* Poor general condition (ASA IV)
* Incomplete colonoscopy planned

Min Age: 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1572 (Estimated)
Dates: Start 2020-10-28 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Adenoma detection rate | during procedure to histological examination result, approximately 2 days
  Difference in adenoma detection rate (all adenomas/all patients) between the two groups

SECONDARY OUTCOMES:
Patient rate difference | during procedure to histological examination result, approximately 2 days
  Differences in the patient rate with adenomas (adenoma detection rate, i.e. rate of patients with at least one adenoma)
Adenoma subgroup differences | histological examination result, approximately 2 days
  Differences subgroups of adenomas (flat, small, high-grade dysplasia)
rate of hyperplastic polyp detection in both groups | histological examination result, approximately 2 days
  Differences in the detection of hyperplastic polyps
rate of polyp detection in preventive and diagnostic colonoscopy | during procedure to histological examination result, approximately 2 days
  Differences in preventive vs. diagnostic colonoscopy
Switching number (BLI, LCI) in both groups | during procedure
  number of switches to visual support by colour filters
incidence of reasons for switching to BLI/LCI | during procedure
  reasons for switching to visual support by colour filters
quality of polyp detection rate by image evaluation | until 2 months after recruitment stop
  differential diagnosis of colon polyps in both groups with/without CADEYE)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Rösch, Prof. dr., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (10):
- Germany (10):
  - Gastroenterologiepraxis Dr. Moog, Kassel, Hesse
  - Universitätsklinikum Leipzig, Leipzig, Saxony
  - GastroZentrum Lippe, Bad Salzuflen
  - Gastroenterologie am Bayerischen Platz, Berlin
  - University Hospital Bonn, Bonn
  - St. Vinzenz-Hospital / Akademisches Lehrkrankenhaus der Universität zu Köln, Cologne
  - University Hospital Eppendorf, Hamburg
  - University Hospital Magdeburg, Magdeburg
  - Marienhospital Osnabrück, Osnabrück
  - Asklepios Paulinen Klinik Wiesbaden, Wiesbaden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Imperiale TF, Glowinski EA, Lin-Cooper C, Larkin GN, Rogge JD, Ransohoff DF. Five-year risk of colorectal neoplasia after negative screening colonoscopy. N Engl J Med. 2008 Sep 18;359(12):1218-24. doi: 10.1056/NEJMoa0803597. PMID 18799558
- [Background] Winawer SJ, Zauber AG, Gerdes H, O'Brien MJ, Gottlieb LS, Sternberg SS, Bond JH, Waye JD, Schapiro M, Panish JF, et al. Risk of colorectal cancer in the families of patients with adenomatous polyps. National Polyp Study Workgroup. N Engl J Med. 1996 Jan 11;334(2):82-7. doi: 10.1056/NEJM199601113340204. PMID 8531963
- [Background] European Colorectal Cancer Screening Guidelines Working Group; von Karsa L, Patnick J, Segnan N, Atkin W, Halloran S, Lansdorp-Vogelaar I, Malila N, Minozzi S, Moss S, Quirke P, Steele RJ, Vieth M, Aabakken L, Altenhofen L, Ancelle-Park R, Antoljak N, Anttila A, Armaroli P, Arrossi S, Austoker J, Banzi R, Bellisario C, Blom J, Brenner H, Bretthauer M, Camargo Cancela M, Costamagna G, Cuzick J, Dai M, Daniel J, Dekker E, Delicata N, Ducarroz S, Erfkamp H, Espinas JA, Faivre J, Faulds Wood L, Flugelman A, Frkovic-Grazio S, Geller B, Giordano L, Grazzini G, Green J, Hamashima C, Herrmann C, Hewitson P, Hoff G, Holten I, Jover R, Kaminski MF, Kuipers EJ, Kurtinaitis J, Lambert R, Launoy G, Lee W, Leicester R, Leja M, Lieberman D, Lignini T, Lucas E, Lynge E, Madai S, Marinho J, Maucec Zakotnik J, Minoli G, Monk C, Morais A, Muwonge R, Nadel M, Neamtiu L, Peris Tuser M, Pignone M, Pox C, Primic-Zakelj M, Psaila J, Rabeneck L, Ransohoff D, Rasmussen M, Regula J, Ren J, Rennert G, Rey J, Riddell RH, Risio M, Rodrigues V, Saito H, Sauvaget C, Scharpantgen A, Schmiegel W, Senore C, Siddiqi M, Sighoko D, Smith R, Smith S, Suchanek S, Suonio E, Tong W, Tornberg S, Van Cutsem E, Vignatelli L, Villain P, Voti L, Watanabe H, Watson J, Winawer S, Young G, Zaksas V, Zappa M, Valori R. European guidelines for quality assurance in colorectal cancer screening and diagnosis: overview and introduction to the full supplement publication. Endoscopy. 2013;45(1):51-9. doi: 10.1055/s-0032-1325997. Epub 2012 Dec 4. PMID 23212726
- [Background] Millan MS, Gross P, Manilich E, Church JM. Adenoma detection rate: the real indicator of quality in colonoscopy. Dis Colon Rectum. 2008 Aug;51(8):1217-20. doi: 10.1007/s10350-008-9315-3. Epub 2008 May 24. PMID 18500502
- [Background] Bretagne JF, Ponchon T. Do we need to embrace adenoma detection rate as the main quality control parameter during colonoscopy? Endoscopy. 2008 Jun;40(6):523-8. doi: 10.1055/s-2007-995786. Epub 2008 May 8. No abstract available. PMID 18464196
- [Background] Corley DA, Jensen CD, Marks AR, Zhao WK, Lee JK, Doubeni CA, Zauber AG, de Boer J, Fireman BH, Schottinger JE, Quinn VP, Ghai NR, Levin TR, Quesenberry CP. Adenoma detection rate and risk of colorectal cancer and death. N Engl J Med. 2014 Apr 3;370(14):1298-306. doi: 10.1056/NEJMoa1309086. PMID 24693890
- [Background] Kaminski MF, Regula J, Kraszewska E, Polkowski M, Wojciechowska U, Didkowska J, Zwierko M, Rupinski M, Nowacki MP, Butruk E. Quality indicators for colonoscopy and the risk of interval cancer. N Engl J Med. 2010 May 13;362(19):1795-803. doi: 10.1056/NEJMoa0907667. PMID 20463339
- [Background] Barclay RL, Vicari JJ, Doughty AS, Johanson JF, Greenlaw RL. Colonoscopic withdrawal times and adenoma detection during screening colonoscopy. N Engl J Med. 2006 Dec 14;355(24):2533-41. doi: 10.1056/NEJMoa055498. PMID 17167136
- [Background] Adler A, Wegscheider K, Lieberman D, Aminalai A, Aschenbeck J, Drossel R, Mayr M, Mross M, Scheel M, Schroder A, Gerber K, Stange G, Roll S, Gauger U, Wiedenmann B, Altenhofen L, Rosch T. Factors determining the quality of screening colonoscopy: a prospective study on adenoma detection rates, from 12,134 examinations (Berlin colonoscopy project 3, BECOP-3). Gut. 2013 Feb;62(2):236-41. doi: 10.1136/gutjnl-2011-300167. Epub 2012 Mar 22. PMID 22442161
- [Background] Adler A, Aminalai A, Aschenbeck J, Drossel R, Mayr M, Scheel M, Schroder A, Yenerim T, Wiedenmann B, Gauger U, Roll S, Rosch T. Latest generation, wide-angle, high-definition colonoscopes increase adenoma detection rate. Clin Gastroenterol Hepatol. 2012 Feb;10(2):155-9. doi: 10.1016/j.cgh.2011.10.026. Epub 2011 Nov 2. PMID 22056301
- [Background] Adler A, Aschenbeck J, Yenerim T, Mayr M, Aminalai A, Drossel R, Schroder A, Scheel M, Wiedenmann B, Rosch T. Narrow-band versus white-light high definition television endoscopic imaging for screening colonoscopy: a prospective randomized trial. Gastroenterology. 2009 Feb;136(2):410-6.e1; quiz 715. doi: 10.1053/j.gastro.2008.10.022. Epub 2008 Oct 15. PMID 19014944
- [Background] Adler A, Pohl H, Papanikolaou IS, Abou-Rebyeh H, Schachschal G, Veltzke-Schlieker W, Khalifa AC, Setka E, Koch M, Wiedenmann B, Rosch T. A prospective randomised study on narrow-band imaging versus conventional colonoscopy for adenoma detection: does narrow-band imaging induce a learning effect? Gut. 2008 Jan;57(1):59-64. doi: 10.1136/gut.2007.123539. Epub 2007 Aug 6. PMID 17681999
- [Background] Adler A, Roll S, Marowski B, Drossel R, Rehs HU, Willich SN, Riese J, Wiedenmann B, Rosch T; Berlin Private-Practice Gastroenterology Working Group. Appropriateness of colonoscopy in the era of colorectal cancer screening: a prospective, multicenter study in a private-practice setting (Berlin Colonoscopy Project 1, BECOP 1). Dis Colon Rectum. 2007 Oct;50(10):1628-38. doi: 10.1007/s10350-007-9029-y. PMID 17694415
- [Background] Schachschal G, Mayr M, Treszl A, Balzer K, Wegscheider K, Aschenbeck J, Aminalai A, Drossel R, Schroder A, Scheel M, Bothe CH, Bruhn JP, Burmeister W, Stange G, Bahr C, Kiesslich R, Rosch T. Endoscopic versus histological characterisation of polyps during screening colonoscopy. Gut. 2014 Mar;63(3):458-65. doi: 10.1136/gutjnl-2013-304562. Epub 2013 Jun 28. PMID 23812324
- [Background] Schachschal G, Sehner S, Choschzick M, Aust D, Brandl L, Vieth M, Wegscheider K, Baretton GB, Kirchner T, Sauter G, Rosch T. Impact of reassessment of colonic hyperplastic polyps by expert GI pathologists. Int J Colorectal Dis. 2016 Mar;31(3):675-83. doi: 10.1007/s00384-016-2523-8. Epub 2016 Feb 4. PMID 26847619
- [Background] Zimmermann-Fraedrich K, Groth S, Sehner S, Schubert S, Aschenbeck J, Mayr M, Aminalai A, Schroder A, Bruhn JP, Blaker M, Rosch T, Schachschal G. Effects of two instrument-generation changes on adenoma detection rate during screening colonoscopy: results from a prospective randomized comparative study. Endoscopy. 2018 Sep;50(9):878-885. doi: 10.1055/a-0607-2636. Epub 2018 Jul 23. PMID 30036893
- [Background] Rosch T, Altenhofen L, Kretschmann J, Hagen B, Brenner H, Pox C, Schmiegel W, Theilmeier A, Aschenbeck J, Tannapfel A, von Stillfried D, Zimmermann-Fraedrich K, Wegscheider K. Risk of Malignancy in Adenomas Detected During Screening Colonoscopy. Clin Gastroenterol Hepatol. 2018 Nov;16(11):1754-1761. doi: 10.1016/j.cgh.2018.05.043. Epub 2018 Jun 11. PMID 29902640
- [Background] Pioche M, Denis A, Allescher HD, Andrisani G, Costamagna G, Dekker E, Fockens P, Gerges C, Groth S, Kandler J, Lienhart I, Neuhaus H, Petruzziello L, Schachschal G, Tytgat K, Wallner J, Weingart V, Touzet S, Ponchon T, Rosch T. Impact of 2 generational improvements in colonoscopes on adenoma miss rates: results of a prospective randomized multicenter tandem study. Gastrointest Endosc. 2018 Jul;88(1):107-116. doi: 10.1016/j.gie.2018.01.025. Epub 2018 Feb 4. PMID 29410020
- [Background] Bronzwaer MES, Dekker E, Weingart V, Groth S, Pioche M, Rivory J, Beyna T, Neuhaus H, Ponchon T, Allescher H, Fockens P, Rosch T. Feasibility, safety, and diagnostic yield of the Extra Wide Angle View (EWAVE) colonoscope for the detection of colorectal lesions. Endoscopy. 2018 Jan;50(1):63-68. doi: 10.1055/s-0043-120666. Epub 2017 Nov 13. PMID 29132174
- [Derived] Zimmermann-Fraedrich K, Sehner S, Rosch T, Aschenbeck J, Schubert S, Liceni T, Moog G, Neumann H, Berndt R, Weigt J, Kaczmarek DJ, May A, Hoffmeister A, Moschler O, Wiessner C, Schachschal G. No Effect of Computer-Aided Diagnosis on Colonoscopic Adenoma Detection in a Large Pragmatic Multicenter Randomized Study. Am J Gastroenterol. 2025 Apr 28. doi: 10.14309/ajg.0000000000003500. Online ahead of print. PMID 40293139